CLINICAL TRIAL: NCT01960114
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Efficacy, Safety, and Pharmacokinetics Study of Extended-Release (ER) Acetaminophen in Postoperative Dental Pain
Brief Title: Study of Long-Acting Acetaminophen in Postoperative Dental Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McNeil Consumer Healthcare Division of McNEIL-PPC, Inc. (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AERPAI2001
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-06

CONDITIONS: Dental Pain
Keywords: Acetaminophen; Paracetamol Analgesics; Analgesics; Non-Narcotic Pain; Postoperative Pain; Antipyretics Dental Surgery; Third molar extraction
MeSH Terms: conditions — Toothache; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen ER (Experimental)
  Interventions: Drug: Acetaminophen ER
- Placebo (Placebo Comparator): Single dose (2 tablets) Acetaminophen ER 750 mg matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen ER — Single dose (2 tablets) Acetaminophen ER 750 mg
  Arms: Acetaminophen ER
Drug: Placebo — Single dose (2 tablets) Acetaminophen ER 750 mg matching placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of acetaminophen ER 1500 mg (two 750 mg tablets) over 10 to 12 hours in the dental pain model following third molar extraction(s) and to evaluate the pharmacokinetics of acetaminophen ER 1500 mg (two 750 mg tablets) in a sub-group of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 17 and less than 46 years of age
* Must weigh at least 100 lbs with a body mass index of at least 18 and less than 30
* Scheduled to undergo surgical extraction of one impacted third molar from the lower jaw. The third molar from the upper jaw from the same side may also be removed.
* Experiencing moderate to severe pain after extraction of third molars.

Exclusion Criteria:

* Cannot be allergic to acetaminophen (Tylenol) or any non-steroidal anti-inflammatory drugs (e.g., Motrin, Advil, Aleve, Naproxen).
* Cannot be pregnant (or planning to be pregnant) or nursing a baby
* Unable to swallow whole large tablets or caplets.
* Cannot have any other medical conditions that the investigator feels may compromise your safety or the study results.

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 403 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Study Director, Study Director — McNeil Consumer Healthcare Division of McNEIL-PPC, Inc.
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (two matching placebo tablets)
- ACE ER 1500 mg: Acetaminophen ER 1500 mg (two 750 mg ER tablets)
Period: Overall Study
Arm/Group | Placebo | ACE ER 1500 mg
Started | 134 | 269
Completed | 133 | 268
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Could not swallow study medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ACE ER 1500 mg | Total
Number analyzed (Participants) | 134 | 269 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.6 (2.66) | 19.5 (2.82) | 19.6 (2.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 143 | 215
  Male | 62 | 126 | 188
Region of Enrollment [Number; unit: participants]
  USA | 134 | 269 | 403

OUTCOME MEASURES:

1. Primary Outcome: Time Weighted Sum of Pain Intensity Difference (PID) Over 10 Hours (SPID 0-10)
Description: Time weighted sum of pain intensity difference scores from baseline over 10 hours. Pain intensity was evaluated using a 0-10 numerical rating scale (NRS) where 0 = no pain and 10 = very severe pain. SPID 0-10 = 0.25 x (PID at 15 min + PID at 30 min + PID at 45 min + PID at 60 min + PID at 75 min + PID at 90 min) + 0.5 x (PID at 120 min) + PID at 3 h + PID at 4 h + PID at 5 h + PID at 6 h + PID at 7 h + PID at 8 h + PID at 9 h + PID at 10 h.
Time Frame: 10 Hours
Population: Analysis was based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ACE ER 1500 mg
Number analyzed (Participants) | 134 | 269
units on a scale | 5.745 (2.5056) | 30.986 (1.8951)
Statistical Analysis 1: Comparison: Placebo vs ACE ER 1500 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical score were factors; Least Squares Mean Difference = 25.241, 95% CI 2-sided [19.669 to 30.813], Standard Error of Mean 2.8344

2. Secondary Outcome: Time to Confirmed First Perceptible Pain Relief
Description: Minutes until confirmed first perceptible pain relief was achieved. Stopwatch was started after the subject took the study medication. The subject was instructed to stop the stopwatch when they first began to feel any pain relief. The first perceptible pain relief was confirmed if the subject also stopped the second stopwatch indicating meaningful pain relief.
Time Frame: Within 12 Hours
Population: Analysis was based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | ACE ER 1500 mg
Number analyzed (Participants) | 134 | 268
Minutes | NA [NA to NA] — Data for the placebo group are not available. Median and 95% Confidence Interval were not estimable because fewer than 50% of the subjects treated with Placebo obtained perceptible pain relief. | 26.817 [23.683 to 29.950]
Statistical Analysis 1: Comparison: Placebo vs ACE ER 1500 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Wilcoxon test, from SAS PROC LIFETEST — The significance threshold level was 0.05 (two-sided). p-Values are based on the Wilcoxon test from PROC LIFETEST that compared survival curves

3. Secondary Outcome: Time to Meaningful Pain Relief
Description: Minutes until meaningful pain relief was achieved. Stopwatch was started after the subject took the study medication. The subjects were instructed to stop the stopwatch when the relief from the starting pain was meaningful to them.
Time Frame: Within 12 Hours
Population: Analysis was based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | ACE ER 1500 mg
Number analyzed (Participants) | 134 | 268
Minutes | NA [NA to NA] — Data for the placebo group are not available. Median and 95% Confidence Interval were not estimable because fewer than 50% of the subjects treated with Placebo obtained meaningful pain relief. | 84.675 [66.333 to 120.633]
Statistical Analysis 1: Comparison: Placebo vs ACE ER 1500 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Wilcoxon test, from SAS PROC LIFETEST — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Duration of Pain Relief
Description: Minutes until rescue medication was given.
Time Frame: Within 12 Hours
Population: Analysis was based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | ACE ER 1500 mg
Number analyzed (Participants) | 134 | 268
Minutes | 106.5 [99.000 to 132.000] | NA [NA to NA] — Data for the acetaminophen ER 1500 mg group are not available. Median and 95% Confidence Interval were not estimable since fewer than 50% of the subjects treated with acetaminophen ER 1500 mg rescued.
Statistical Analysis 1: Comparison: Placebo vs ACE ER 1500 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups. Subjects who withdrew from the study before 12 hours, but did not use rescue therapy, were censored at the time of withdrawal. Subjects not rescuing during the 12-hour study period had their time to rescue set to 12 hours and were censored; Test type: Superiority or Other; p < 0.001, Log Rank — The significance threshold level was 0.05 (two-sided). p-Values are based on the log-rank test from PROC LIFETEST that compared survival curves

5. Secondary Outcome: Patient Global Evaluation
Description: Patient Assessment of the pain medication - Number of subjects rating the medication they received as a pain reliever on a score of 0-4, where 0=poor, 1=fair, 2=good, 3=very good, 4=excellent.
Time Frame: 12 Hours
Population: Analysis was based on the Intent-to-Treat (ITT) population, which included all subjects who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | ACE ER 1500 mg
Number analyzed (Participants) | 133 | 268
percentage of participants
  Poor (0) | 63.2 | 18.3
  Fair (1) | 9.0 | 11.2
  Good (2) | 8.3 | 14.6
  Very Good (3) | 12.8 | 35.8
  Excellent (4) | 6.8 | 20.1
Statistical Analysis 1: Comparison: Placebo vs ACE ER 1500 mg; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); Used row-mean scores based on Cochran-Mantel-Haenszel test was stratified by baseline categorical pain score

ADVERSE EVENTS:
Time Frame: Day 5-7 for non-serious adverse events, until 30 days after the last study site visit for serious adverse events.
Description: Adverse events were systematically collected at each study visit through the Follow Up Telephone Call (Day 5-7). Serious adverse events were reported through 30 days after the participant's last study site visit. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | Placebo | ACE ER 1500 mg
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/268
Other Adverse Events (participants affected / at risk) | 14/134 | 26/268
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=134) | ACE ER 1500 mg (N=268)
Nausea (Gastrointestinal disorders) | 14 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less